CLINICAL TRIAL: NCT04263519
Title: A Pilot Open Labeled Study of Tacrolimus to Assess it's Effects on Bio-markers of Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: A Pilot Open Labeled Study of Tacrolimus in Alzheimer's Disease.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid restrictions
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven E Arnold, Manager Director Phsycian, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003904
Record Dates: First submitted 2020-01-23; First posted 2020-02-10 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Serum Level (Active Comparator): Stable Blood Tacrolimus of 2-5 ng/ml.
  Interventions: Drug: Tacrolimus
- High Serum Level (Active Comparator): Stable Blood Tacrolimus of 5.1-10 ng/ml.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Oral Immunosuppressant

SUMMARY:
A Pilot open labeled study of Tacrolimus in Alzheimer's Disease.

DETAILED DESCRIPTION:
This study will investigate the neurobiological effect of tacrolimus in persons with MCI and dementia due to AD by measuring biomarkers of target engagement in immune response, amyloid-b, tau and neurodegeneration in CSF, functional connectivity with MRI and EEG, and cognition. Study objectives include:

ELIGIBILITY:
Inclusion Criteria:

Study subjects meeting all of the following criteria will be allowed to enroll in the study:

1. Age 55-85 inclusive, male or female.
2. Diagnosis of MCI or dementia due to AD as shown by positive AD biomarker (CSF or neuroimaging).
3. Education level, English language skills and literacy indicates subject will be able to complete all assessments.
4. Willing and able to complete all assessment and study procedures, including phlebotomies, lumbar punctures, MRIs, neurocognitive testing.
5. Subject has a study partner with at least two days of contact per week and willingness to assist with subject's research activities.
6. If on cholinesterase inhibitor and/or memantine, doses are stable for 3 months prior to baseline.

Exclusion Criteria:

Subjects meeting any of the following criteria during the screening evaluation will be excluded:

1. Allergy or hypersensitivity to tacrolimus.
2. Any specific CNS disease other than suspected AD, such as major clinical stroke, brain tumor, normal pressure hydrocephalus, multiple sclerosis, significant head trauma with persistent neurological of cognitive deficits or complaints, Parkinson's disease, frontotemporal dementia, and/or other neurodegenerative diseases.
3. Any significant systemic illness or clinically significant unstable medical condition that could affect subject safety or compliance with the study; including but not limited to any active infection, active malignancy except non-melanomatous skin cancers, cirrhosis, active hepatitis, uncontrolled diabetes (A1c >8), AIDS, common variable immunodeficiency, conditions treated with biologics, uncontrolled hypertension, chronic kidney disease with an eGFR <45 ml/min, Platelets < 100K, Hgb <9.
4. History of alcohol or other substance abuse or dependence with the past two years.
5. Major active psychiatric illness (e.g. depression, bipolar disorder, obsessive compulsive disorder, schizophrenia) within the previous year.
6. Current suicidal ideation or history of suicide attempt.
7. Contraindications to undergo MRI studies:

   1. History of a cardiac pacemaker or pacemaker wires,
   2. Metallic particles in the body,
   3. Vascular clips in the head,
   4. Prosthetic heart valves, or
   5. Severe claustrophobia impeding ability to participate in an imaging study.
8. MRI findings that show one or more of the following:

   1. More than 4 incidental microhemorrhages,
   2. Incidental lacunar infarcts with attributable signs or symptoms and with history of stroke,
   3. Incidental meningiomas with attributable signs or symptoms, or
   4. Newly recognized meningioma.
9. Laboratory abnormalities in B12, TSH, or other common laboratory parameters that may contribute to cognitive dysfunction.
10. Laboratory abnormalities in PT-INR, CBC, electrolytes, magnesium, LFTs, BUN, Cr or others, or abnormalities in ECG posing risk to treatment with tacrolimus.
11. Current use of medications with psychoactive properties (e.g., anticholinergics, antihistamines, antipsychotics, sedative hypnotics, anxiolytics) that may deleteriously affect cognition in the judgement of the investigator.
12. Current use of medications that interact with tacrolimus (protease inhibitors, macrolides, rifampin, barbiturates, phenytoin, or azoles).
13. Inability to avoid any dietary supplements that could interact with tacrolimus metabolism.
14. Inability to avoid grapefruit and grapefruit juice.
15. Use of other small molecule or device-based investigational agents one month prior to entry and for the duration of the trial; or participation in any immunotherapy clinical trial within three months prior to baseline visit.
16. Discontinuation of cholinesterase inhibitor or memantine within one month (28 days) prior to baseline visit.
17. Females who are pregnant, lactating or of child-bearing potential

    -

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
CSF biomarkers of target engagement, AD pathology, and neurodegeneration | Baseline and 12 weeks
  Evaluate effect of tacrolimus on molecular markers of target engagement (calcineurin/NFAT mediated inflammatory markers IL-2, IL-6, IFNβ and YKL-40), AD pathology (amyloid-β, tau, phospho-tau) and neurodegeneration (neurofilament-light, neurogranin). We will measure change from baseline in all CSF biomarkers following 12 weeks of steady treatment.

SECONDARY OUTCOMES:
Blood biomarkers of target engagement, AD pathology, and neurodegeneration. | Baseline and 12 weeks
  Evaluate effect of tacrolimus on molecular markers of target engagement (calcineurin/NFAT mediated inflammatory markers IL-2, IL-6, IFNβ and YKL-40), AD pathology (amyloid-β, tau, phospho-tau) and neurodegeneration (neurofilament-light, neurogranin). We will measure change from baseline in all blood biomarkers following 12 weeks of steady treatment.
Structural neuroimaging of Hippocampal volume. | Baseline and 12 weeks
  Evaluate effect of tacrolimus on size of different brain regions using Magnetic Resonance Imaging (MRI). We will measure change from baseline after 12 weeks of treatment.
Functional neuroimaging of default mode network connectivity. | Baseline and 12 weeks
  Evaluate effect of tacrolimus on blood flow to different brain regions using functional MRI (fMRI). We will measure change from baseline after 12 weeks of treatment.
Electroencephalograms (EEG) spectral power | Baseline and 12 weeks
  Evaluate effect of tacrolimus on resting state EEG frequency using the linear power spectral density technique. We will measure change from baseline after 12 weeks of treatment.
Montreal Cognitive Assessment (MoCA) | Baseline and 12 weeks
  Evaluate effect of tacrolimus on major domains of cognition (score range 0-30, high is better). We will measure change from baseline after 12 weeks of treatment.
Neuropsychiatric Inventory Questionnaire (NPIQ) | Baseline, 4 weeks, 8 weeks and 12 weeks
  Evaluate effect of tacrolimus on neuropsychiatric symptoms as rated by a study partner/informant (score range 0-80, high is worse). We will measure change from baseline after 4, 8, and 12 weeks of treatment.
Functional Activities Questionnaire (FAQ) | Baseline, 4 weeks, 8 weeks and 12 weeks
  Evaluate effect of tacrolimus on ability to daily functional ability as reported by study partner/informant (score range (0-30, low is better). We will measure change from baseline after 4, 8, and 12 weeks of treatment.
Repeated Battery for the Assessment of Neuropsychological Status | Baseline, 4 weeks, 8 weeks and 12 weeks
  Evaluate the effect of tacrolimus on several domains of cognitive function (score range 40-160, higher is better). We will measure change from baseline after 4, 8, and 12 weeks of treatment.

IPD SHARING:
Plan to Share IPD: No